CLINICAL TRIAL: NCT03794388
Title: Multicentric, Open, Randomized Study Comparing Topical Treatment by Patch of Capsaicin to 8% (Qutenza) to Pregabalin Oral in the Early Treatment of Neuropathic Pain After Primary Surgery for Breast Cancer
Brief Title: Evaluation in the Treatment of Neuropathic Pain Post Breast Surgery
Acronym: CAPTRANE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ICO-A-2018-10
Record Dates: First submitted 2018-11-05; First posted 2019-01-07 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer Patient
Keywords: Breast cancer patient; Surgery; Inter Costobrachial Neuralgia
MeSH Terms: interventions — Capsaicin; Pregabalin

STUDY DESIGN:
Intervention Model Description: Multicenter, open, randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm CAPSAICINE topical (Experimental): Application of capsaicin patches at 8% on the painful area
  1 to 2 patches will be administered during the consultation. If necessary, a second application will be realized 3 months later.
  Interventions: Drug: Capsaicin
- Arm PREGABALINE (Active Comparator): Pregabalin tablets will be initiated at a dose of 50 mg / day taken in 2 doses Depending on the tolerance, the dose will be increased to 100 mg / day and then to 150 mg / day to reach a maximum dose of 600 mg / day.
  An interval of 3 to 7 days must be observed between each dose increase.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Capsaicin — Application of capsaicin patches at 8% on painful area
  Other Names: qutenza EU/1/09/524/001
  Arms: Arm CAPSAICINE topical
Drug: Pregabalin — Taking Pregabalin tablets
  Other Names: Lyrica
  Arms: Arm PREGABALINE

SUMMARY:
Breast cancer is the most common cancer in women in Europe. Therefore, breast cancer has become a chronic disease and patients need to learn to live with it as well as with the adverse effects related to the disease itself or to the therapies used.

As noted in the third "Plan cancer", pain is a major criterion in the quality of life of patients treated for breast cancer.

Neuropathic pain was defined in 2011 by the international Association for the Study of Pain (I.A.S.P.) as the direct result of a lesion or disease affecting the somato-sensory system.

Surgical treatment is often the first treatment of breast cancer. It can be conservative by performing a partial mastectomy (lumpectomy or quadrantectomy) or non-preservative by total mastectomy.

Intercostobrachial neuralgia (NICB) or Post mastectomy painful Syndrome (MPRR) was first described by Wood in 1978 as "chronic pain beginning immediately or early after a mastectomy" Or a lumpectomy affecting the anterior thorax, armpit and/or arm in its upper half. These post-surgical pains are related to a lesion of the nerves in the breast area.

In particular, the intercostobrachial nerve can be severed, stretched or crushed during surgery.

Post-operative neuropathic pain in patients with breast cancer is underdiagnosed either by general practitioner or in a specialized environment.

The diagnosis of neuropathic pain is performed during examination and clinical examination. Several scales allow to detect neuropathic pain but only the DN4 is recognized to be the most specific and sensitive scale.

Patients do not always express this pain. They do not always reconcile with the surgery. Either because the pain occurs a long time after the surgery, or they find it normal to get hurt. These diagnostic difficulties cause a delay in setting up a suitable analgesic treatment.

However, neuropathic pain responds poorly to common analgesics. Diagnosis, evaluation and early management of neuropathic pain are a priority in order to avoid their chronicization, to improve the quality of life of patients with breast cancer and to enable them to return to work quickly.

We therefore assume that the diagnosis of early neuropathic pain at 2 months of surgery associated with initiation of appropriate topical treatment without the systemic effects of conventional oral treatments, would reduce the incidence of Chronic neuropathic pain 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female who had first breast cancer surgery, regardless of the type of surgery
* Age ≥ 18 years
* Healthy, non-irritated skin on painful areas to treat
* During the inclusion visit to M4 post surgery, neuropathic pain of the breast and / or axillary area corresponding to inter-brachial neuralgia with a DN4≥4 score.
* Obtaining the signed written consent of the patient
* Major patient affiliated to a social security scheme

Exclusion Criteria:

* Contraindications specific to the treatments studied : capsaicine and pregabalin
* Diabetic patient
* Previous treatment with capsaicin or pregabalin
* Opioid treatment> 80 mg / day (oral morphine equivalent) in progress- Topical treatment of pain between surgery and inclusion visit
* Uncontrolled hypertension (systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 90 mmHg) or recent history (<3 months) of cardiovascular events (stroke, heart attack, pulmonary embolism)
* Creatinine clearance (CLcr) <60mL / min according to the Cockcroft-Gault formula
* Pregnant woman, likely to be pregnant or breastfeeding
* Persons deprived of their liberty or guardianship (including curators),
* Impossibility of submitting to the medical follow-up of the test for geographical, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
To show the noninferiority of early early medical treatment by topical treatment with capsaicin compared to oral treatment of pregabalin on the evolution of neuropathic pain after 2 months in patients who have undergone surgical excision of breast cancer | 2 months
  The 11-point numerical scale (0-10) is collected at 2 months.

SECONDARY OUTCOMES:
To compare the efficacy of an early medical treatment with capsaicin topical treatment compared to oral treatment pregabalin on the evolution of neuropathic pain in patients who had undergone excision surgical breast cancer after 6 months of treatment | 6 months
  The 11-point numerical scale of pain is also collected at the end of treatment
To compare the functional change and quality of life perceived by patients after 2 and 6 months of treatment between the two arms: Questionnaire PGIC (patients' global impression of change) | 6 months
  Questionnaire PGIC is administered to M4, M6 and at the end of treatment to measure the functional changes and quality of life changes experienced by the patient in the 2 treatment arms.
To compare the functional change and quality of life perceived by patients after 2 and 6 months of treatment between the two arms | 6 months
  Questionnaire QLQ-C30 (quality of life questionnaire) is administered to M4, M6 and at the end of treatment to measure the functional changes and quality of life changes experienced by the patient in the 2 treatment arms.
To compare the functional change and quality of life perceived by patients after 2 and 6 months of treatment between the two arms | 6 months
  Questionnaire EQ-5D is administered to M4, M6 and at the end of treatment to measure the functional changes and quality of life changes experienced by the patient in the 2 treatment arms.
Regression of the painful area after 2 and 6 months of treatment between the two arms. | 6 months
  The painful area is measured from pain mapping at baseline, and after 2 months and 6 months of treatment. It is measured by the area delimited by the contours of the painful surface (centralized reading).
Tolerance of each type of treatment by collecting side effects in each treatment arm. | 6 months
  The tolerance of the treatments will be measured by the number of patients having at least one adverse event of grade ≥ 2 according to the classification CTCAE v5.0.
Proportion of patients for whom only 1 application has been sufficient. | 6 months
  In the capsaicin arm, the number of total patches received by the patient during the 6 months will also be counted
Impact of peri-surgical anxiety and depression on the development of neuropathic pain after surgery for breast cancer | 49 months
  The HAD (Hospital anxiety and despression scale) questionnaire will be collected during the screening visit
The incidence of NICBs 4 months after surgery for breast cancer | 4 months
  The incidence of NICBs will be measured by the number of patients included in the study (DN4 +) compared to the number of patients screened before surgery
The evolution of the weight between the two arms after 6 months of treatment. | 6 months
  The weight is collected after 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: DENIS DUPOIRON, MD, Study Director — Institut de Cancérologie de l'Ouest
Locations (11):
- France (11):
  - Institut de Cancerologie de L'Ouest, Angers
  - Chu Grenoble, Grenoble
  - Chd Vendee, La Roche-sur-Yon
  - Centre Oscar Lambret, Lille
  - Hopital Saint Vincent de Paul, Lille
  - Centre Leon Berard, Lyon
  - CHU NICE, Nice
  - Institut Jean Godinot, Reims
  - Institut Curie, Saint-Cloud
  - Iuct Oncopole, Toulouse
  - Ch Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No